CLINICAL TRIAL: NCT02868788
Title: Anti-inflammatory and Reactive Oxygen Species (ROS) Suppressive Effects of the Fiber Supplementation to a High Fat High Carbohydrate Meal and Fiber Supplementation Alone in Obese Patients With Type 2 Diabetes
Brief Title: Anti-inflammatory Effects of the Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, SUNY Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1977
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
Keywords: inflammation; insulin resistance; type 2 diabetes; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Insulin Resistance; Obesity | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high fat high calorie meal (HFHC) (Other): Subjects in this arm will receive high fat high calorie (HFHC) meal only
  Interventions: Other: HFHC meal
- HFHC plus fiber (Experimental): Subjects in this arm will receive HFHC meal plus dietary fiber supplementation
  Interventions: Dietary Supplement: dietary fiber; Other: HFHC meal

INTERVENTIONS:
Dietary Supplement: dietary fiber — Fiber one supplement (32 grams of fiber) will be consumed with 910 Calorie HFHC meal
  Other Names: Fiber One
  Arms: HFHC plus fiber
Other: HFHC meal — 910 Calorie HFHC meal

SUMMARY:
This study will help elucidate the mechanism underlying the cardioprotective and anti-diabetes effect of dietary fiber by exploring a comprehensive set of inflammatory and oxidative stress markers, based on a contemporary understanding of this process. In addition, there have been very few studies that explored the immediate change in oxidative stress and incretin secretion after fiber intake. In this study, the investigators will be able assess the short term metabolic impact of dietary fiber at great details. The result will contribute to dietary recommendation or designing of fiber supplementation for prevention/treatment of diabetes, obesity and cardiovascular disease.

DETAILED DESCRIPTION:
Baseline labs include complete blood count (CBC), comprehensive metabolic panel (CMP), Hemoglobin A1C, and lipid profile. All labs will be drawn in the fasting state

Visit 1: Subjects will arrive after having fasted overnight (10 hours) at 7 to 7:30 am. An indwelling intravenous cannula will be placed in the anterior cubital vein for blood draws. A blood sample of the research labs and a urine sample will be collected. Blood pressure, heart rate and weight will be measured. Subjects will consume either a High Fat High Calorie (HFHC) meal or HFHC meal plus fiber (FiberOne Original cereal) according to randomization. Fiber will be consumed before and after the HFHC meal (28 grams in total, 14 grams before and after the meal). HFHC meal includes an egg muffin sandwich, a sausage muffin sandwich and two hash browns which contain 88g carbohydrate, 51 g fat (33% saturated) and 34 g protein. 35 ml of blood will be obtained at 1h , 2h, 3h and 5 h and 5 ml at 15 min,30 min,45 min,75 min and 90 min. A total of 165 ml (11 tablespoon) blood will be collected.

. Visit 2: Subjects will return 1 week later after overnight fasting (10 hours) at 7 to 7:30 am. Blood pressure, heart rate and weight will be measured. Baseline blood and urine samples will be collected again and subjects will be crossed over to receive the second meal (HFHC only or HFHC with fiber). Visit details are similar to visit 1. After this, the subject will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 to 80 years of age
2. Non-smoker (last cigarette at least one month ago)
3. Type 2 diabetes for at least 1 year
4. Body mass index > 30 kg/m2

Exclusion Criteria:

1. Participation in any other concurrent clinical trials
2. Pregnancy or premenopausal women who are trying to be pregnant
3. Patients who are incompetent to give consent
4. Patients on non-steroidal anti-inflammatory drugs or steroids
5. Concurrent disease that could disrupt intestinal epithelium and increase permeability to endotoxin, ie Celiac and Crohns disease.
6. Hepatic disease (transaminase > 3 times normal)
7. Renal impairment (serum creatinine > 1.5 mg/dl)
8. History of drug or alcohol abuse
9. Use of over the counter or prescribed probiotic supplements.
10. Recent or current antibiotic use.
11. Coronary artery disease (CAD): documented by history of myocardial infarction, angioplasty/stent placement, angina, exercise EKG positive for ischemia or angiographic evidence of CAD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HFHC Meal Only First Then HFHC Meal Plus Fiber Second: Subjects in this arm will receive high fat high calorie (HFHC) meal first Then after 1 week will receive HFHC meal Plus Fiber
- HFHC Meal Plus Fiber First Then HFHC Meal Only Second: Subjects in this arm will receive high fat high calorie (HFHC) meal Plus Fiber first Then after 1 week will receive HFHC meal only
Period: First Visit
Arm/Group | HFHC Meal Only First Then HFHC Meal Plus Fiber Second | HFHC Meal Plus Fiber First Then HFHC Meal Only Second
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Visit (One Week Later)
Arm/Group | HFHC Meal Only First Then HFHC Meal Plus Fiber Second | HFHC Meal Plus Fiber First Then HFHC Meal Only Second
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: CROSS-OVER STUDY. So, baseline information for both intervention groups is same
Groups:
- Overall Study Participants: All participants will randomly receive HFHC meal with or without dietary fiber supplementation in first visit and the other intervention in the second visit. Total 10 participants in cross-over design study
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 34 (4)

OUTCOME MEASURES:

1. Primary Outcome: Peak Change in From Baseline in Reactive Oxygen Species (ROS) Generation
Description: mononuclear cells will be isolated by Ficoll-Hypaque method and ROS will be measured by chemiluminescence as an index of NADPH oxidase activation. Measurment will take place at baseline before the meal intervention and hourly for 5 hrs after the meal. The percent change from baseline at peak effect will be calculated.
Time Frame: 5hr
Measure: Mean (Standard Error); unit: percentage of change
Groups:
- High Fat High Calorie: Subjects in this arm will receive high fat high calorie meal
  dietary fiber
- High Fat High Calorie Plus Fiber: Subjects in this arm will receive high fat high calorie meal plus dietary fiber supplementation
  dietary fiber
Arm/Group | High Fat High Calorie | High Fat High Calorie Plus Fiber
Number analyzed (Participants) | 10 | 10
percentage of change | 224 (15) | 167 (13)

2. Secondary Outcome: Peak Change in From Baseline in Nuclear Factor-Kappa B (NFkB) Activation
Description: Nuclear factor-Kappa B (NFkB) activation will be measured at baseline before the meal and hourly up to 5 hrs and percent change from baseline at peak effect is calculated
Time Frame: 5hr
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | High Fat High Calorie | High Fat High Calorie Plus Fiber
Number analyzed (Participants) | 10 | 10
percentage of change | 124 (14) | 109 (8)

3. Secondary Outcome: Percent Change Toll Like Receptor-4 (TLR-4) Levels
Description: Toll Like Receptor-4 will be measured by Western Blots at baseline before meal intake and hourly up to 5 hrs after meal. Percent change from baseline at peak effect is calculated.
Time Frame: 5hr
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | High Fat High Calorie | High Fat High Calorie Plus Fiber
Number analyzed (Participants) | 10 | 10
percentage of change | 181 (15) | 135 (12)

4. Secondary Outcome: Change in Plasma Lipopolysaccharides Level From Baseline.
Description: Lipopolysaccharide will be measured by commercially available kit (Cambrex Limulus Amebocyte Lysate kit, Lonza Inc. Walkersville, MD). Measurements will take place at baseline before the meals and hourly for next 5 hrs. Percent change from baseline at peak effect is calculated.
Time Frame: 5hr
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | High Fat High Calorie | High Fat High Calorie Plus Fiber
Number analyzed (Participants) | 10 | 10
percentage of change | 124 (10) | 128 (11)

ADVERSE EVENTS:
Time Frame: 5hr
Arm/Group | High Fat High Calorie | High Fat High Calorie Plus Fiber
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT02868788/Prot_SAP_000.pdf